CLINICAL TRIAL: NCT02709447
Title: Dating Violence Prevention for Juvenile Justice Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 500421
Record Dates: First submitted 2016-02-09; First posted 2016-03-16 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2020-03

CONDITIONS: Violence
Keywords: Intimate Partner Violence; Juvenile Delinquency; Sexual Behavior
MeSH Terms: conditions — Sexual Behavior | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Date SMART (Experimental): Group based prevention
  Interventions: Behavioral: Date SMART
- Health Promotion (Active Comparator): Group based prevention
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Behavioral: Date SMART — Skills-based, group prevention program targeting emotion regulation and interpersonal skills using a cognitive-behavioral framework.
  Arms: Date SMART
Behavioral: Health Promotion — Psycho-educational group prevention program targeting knowledge and skills only
  Arms: Health Promotion

SUMMARY:
Girls in the juvenile justice system are at high risk for dating violence exposure as well as co-occurring problems with delinquency and sexual risk taking. Despite the multitude of negative outcomes associated with dating violence, no evidence-based preventive interventions exist for juvenile justice girls. This study will advance scientific knowledge by testing the efficacy of a promising, skills-based intervention (Date SMART) on reducing dating violence, delinquency and sexual risk outcomes for a broad range of court-involved, non-incarcerated girls.

DETAILED DESCRIPTION:
Research is urgently needed to rigorously test a skills-based intervention for dating violence prevention among juvenile justice girls. Court-involved, non-incarcerated (CINI) girls represent a particularly high-risk group for dating violence exposure. This is due to the multiple risk factors they possess that have demonstrated associations with teen dating violence outcomes in other high-risk adolescent female populations. Despite the critical need for these young women to learn strategies that offset their heightened risk for involvement in coercive romantic relationships, no such evidence-based interventions exist for this population. The goal of the current study is to establish the efficacy of Date SMART (K23MH086328), a theoretically-driven skills-based intervention, in reducing dating violence, sexual risk behavior, and delinquency among girls in the juvenile justice system. Pilot data reveal that girls randomized to the Date SMART intervention spend significantly fewer days in violent relationships compared to girls randomized to the comparison condition. They also show improvements in condom use at last sex and reductions in delinquency. Moreover, the risk profile of adolescent girls who participated in the pilot trial is remarkably similar to the profile of adolescent girls involved in the juvenile justice system. Thus, Date SMART is uniquely suited for CINI girls. Despite the promise of Date SMART, the time lag from pilot testing to efficacy testing and final dissemination activities is protracted, as researchers fail to consider questions of effectiveness early on. Hybrid designs that retain core components of efficacy trials (randomization, controlled conditions) and essential elements of effectiveness research (e.g., participant diversity; standardized training procedures, attention to cost) can reduce time to implementation in the "real world." As such, investigators plan to test the efficacy of Date SMART on dating violence, sexual risk, and delinquency among 250 court-involved, non-incarcerated girls. Investigators will also gather effectiveness data from key stakeholders to determine how best to implement the program, train staff, and predict the cost of the program within the juvenile court. CINI girls, ages 14-17 (N= 12 juveniles for Phase I Intervention Run-Through; N=250 for Phase II Randomized Control Trial [RCT] study) will be recruited from the Rhode Island Family Court and Probation Departments and randomized to either the Date SMART (active) intervention (n=125) or a Health Promotion (control) condition (n=125). In Phase I (12 juveniles will be recruited to complete the Intervention Run-Through and research assessment once to allow testing of RCT intervention and assessment procedures prior to the RCT phase. In Phase II, 250 juveniles will be recruited and randomized at baseline and then re-assessed at 3, 6, 9 and 12 month post-intervention follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Court-involved, non-incarcerated adolescent female
* Parent/ guardian consent and teen assent

Exclusion Criteria:

* Outside of 14-18 age range
* Cognitive/ developmental delays or psychosis that would interfere with study participation

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 253 (Actual)
Dates: Start 2015-04; Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Dating Violence Perpetration and Victimization from Baseline to 3 months | Baseline and 3 months
  Conflict in Adolescent Dating Relationships Inventory (CADRI) assesses abuse perpetration and victimization with a current or recent dating partner. The CADRI has strong internal consistency (total α = .83) and 2-week test retest reliability, r = .68, p < .01, as well as acceptable partner agreement (r = .64, p < .01) on the basis of 35 couples. At baseline, participants will be asked about the prevalence of DV over the lifetime and the past 3 months. For all other time points, we will assess the past 3 months.

SECONDARY OUTCOMES:
Recidivism over 3 months | Baseline and 3 months
  Juveniles' recidivism rates, description of related charges (e.g., substance-related, property) and time detained/incarcerated (all tracked by the court database) will be available to the project and assessed at baseline and follow-ups.
Change in Unprotected Sex Acts from Baseline to 3 months | Baseline and 3 months
  The Adolescent Risk Behavior Assessment (ARBA) assesses type of sexual behavior, frequency of sex and condom use, number of partners and substance use preceding and/or during sex. Intentions to have sex, use condoms and get pregnant are measured within the ARBA and will be recorded.
Change in Delinquent Behavior from Baseline to 3 months | Baseline and 3 months
  The National Youth Survey Self Reported Delinquency Scale will also be administered and is a self-report of delinquent acts (e.g., larceny, fighting, selling drugs, etc.), the number of times alcohol/drugs were involved in each delinquent act, and number of times the delinquent act was committed to gain access to alcohol/drugs.
Change in Physical and Sexual Dating Violence Perpetration from Baseline to 3 months | Baseline and 3 months
  Timeline Follow-back Spousal Violence Interview (TLFB -SV), adapted for adolescents (and used successfully in pilot trial) assesses the number of days with a dating partner, presence of physical or sexual DV (perpetration or victimization) by day, and presence of alcohol/drug use.

OTHER OUTCOMES:
Change in Depression Symptoms from Baseline to 3 months | Baseline and 3 months
  The Beck Depression Inventory-II (BDI-II) consists of 21 items to assess the intensity of depression. Each item is a list of four statements in increasing severity about a symptom of depression.
Change in Emotion Regulation Skills from Baseline to 3 months | Baseline and 3 months
  The Adolescent Self-Regulatory Inventory (ASRI) is a 33 item survey that measures adolescents' use of both functional and dysfunctional emotion regulation strategies.
Change in Anger Expression from Baseline to 3 months | Baseline and 3 months
  The Anger Expression Scale (AES) of the State-Trait Anger Expression Inventory (STAXI-2) measures control of expressed anger and internal/external anger expression (reliability is good; α's range.73 - .84).

CONTACTS AND LOCATIONS:
Overall Officials: Christie Rizzo, PhD, Principal Investigator — Northeastern University
Locations (1):
- Rhode Island Family Court, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No